CLINICAL TRIAL: NCT04240262
Title: Prospective Observational Trial of Microwave Ablation for Leiomyoma (MYOMIC2)
Brief Title: Microwave Ablation for Leiomyoma
Acronym: MYOMIC2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Senior consultant ob/gyn, Karolinska Institutet
Other Study IDs: MYOMIC2
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate the effectiveness and acceptability of percutaneous or vaginal ultrasound guided microwave ablation for the treatment of symptoms related to uterine fibroids. We will include 200 women.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal
* no future child wish
* acceptable risks for general anestesia or sedation
* willing to comply with protocol

Exclusion Criteria:

* current or future child wish
* bleeding disorder with increased risk of bleeding

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with symptoms from uterine fibroids
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Symptom severity of uterine fibroids | 6 months post treatment
  Score of validated form Uterine Fibroid symptom- Quality of Life questionnaire. minumum 0, maximum 100 where higher scores indicate higher symptom severity

SECONDARY OUTCOMES:
Quality of Life score | 6 months post treatment
  Score of validated form Uterine Fibroid symptom- Quality of Life questionnaire.minumum 0, maximum 100 where higher scores indicate higher quality of life
menstrual bleeding | 6 months post treatment
  Score on validated Pictorial Bleeding assessment chart. minimum 1, no maximum. higher scores indicate more bleeding.
acceptability | 2 hours post treatment and 6 months post treatment (+/- 2 weeks)
  Answer to question: if you were to recommend the treatment to a friend on a scale from 1-7 where 7 is the highest rating- what would you say.

CONTACTS AND LOCATIONS:
Locations (1):
- Helena Kopp Kallner, Täby, Sweden

REFERENCES:
- [Derived] Jonsdottir G, Beermann M, Lanz E, Nikodell A, Cronsioe A, Hasselrot K, Kopp-Kallner H. Ultrasound guided microwave ablation treatment of uterine fibroids: Clinical response and patient acceptability. Acta Obstet Gynecol Scand. 2025 Feb;104(2):350-356. doi: 10.1111/aogs.15041. Epub 2024 Dec 19. PMID 39697096